CLINICAL TRIAL: NCT02617342
Title: Robot-Mediated Social Skills Intervention for Children With Autism Spectrum Disorders
Brief Title: Robot-Mediated Intervention for Children With Autism Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Aetna, Inc. (Industry)
Responsible Party: Principal Investigator, Rebecca Landa, Director of the Center for Autism and Related Disorders (CARD) and Professor, Johns Hopkins, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00067744
Record Dates: First submitted 2015-11-24; First posted 2015-11-30 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder
Keywords: Intervention; Autism Spectrum Disorder; Social Skills
MeSH Terms: conditions — Autism Spectrum Disorder; Social Skills

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robot-mediated Intervention (Experimental): Families assigned to the robot condition will be asked to complete pre-test assessments and post testing as well as to participate in the robot intervention. The intervention will last for a 8-14 week period in which families will bring their child in 2-3 times a week on average for approximately 30 minutes until 24 treatment sessions have been completed. Children will receive one-on-one intervention with an interventionist facilitating the child's interactions with the robot.
  Interventions: Behavioral: Robot-mediated Intervention
- Treatment as Usual (No Intervention): Families assigned to the TAU condition will be asked to complete pre-test assessments and approximately 8-14 weeks later return to complete post-test assessments where the social emotions activity will be retested. During the 8-14 weeks between the testing assessments, families in the TAU condition will also receive a weekly email asking about their child's media use.

INTERVENTIONS:
Behavioral: Robot-mediated Intervention — The intervention follows the curriculum developed by RoboKind to target and improve upon social interactions through core vocabulary and modeling.
  Arms: Robot-mediated Intervention

SUMMARY:
This study is being done to examine the impact of an interactive, social robotics program in helping children with autism spectrum disorders (ASD) understand emotions and how to better recognize emotions while interacting with others. Eligible families will be randomized to either the robot intervention (n=20) or a no intervention (TAU; n=20) condition for 8-14 weeks. Assessments will occur at pre- and post-intervention as well as weekly for both conditions.

ELIGIBILITY:
Inclusion Criteria:

* Child participants must be between the ages of 4 years, 0 months and 8 years, 11 months.
* Children must meet criteria for ASD or autism on the Autism Diagnostic Observation Schedule (ADOS-2; Lord et al., 2012) plus receive a clinical judgment of pervasive developmental disorder not otherwise specified (PDD-NOS) or autism by the study team.
* Children must possess sufficient expressive language skills to qualify for at least an ADOS-2 Module 2.
* Caregivers must agree to participate in the study and commit to having their child participating in the intervention to which they are randomized for approximately three months.
* Caregivers must agree to bring their child in for pre-testing and post-testing.
* Family must speak English at least 50% in the home.

Exclusion Criteria:

* Child IQ <70 (per Stanford Binet short form).
* History of head injury, seizure disorder, severe aggression or self-injurious behavior.
* Vision impairment after correction.
* Cannot be living in foster care.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2015-11; Primary Completion 2017-12-17 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Change in baseline emotions accurately identified on the Transporters Quiz | 14 weeks into treatment (at completion of intervention)
  The Transporters Quiz (Autism Transporters CIC, Autism Research Center) is a quiz developed to test a child's understanding of the emotions portrayed in stories. The quiz examines whether a child can link a word describing an emotion, the facial expression of that emotion, and the causes of the emotion. This quiz will be given prior to starting treatment and again at the completion of the intervention.

SECONDARY OUTCOMES:
Change in baseline Social Responsiveness Scale Score | 14 weeks into treatment (at completion of intervention)
Number of prompt-free intervals during the treatment sessions | Weekly throughout intervention schedule (8-14 weeks)
  For treatment condition only. One session a week will be randomly selected to be recorded for 15 minutes and coded for the number of times the child independently and appropriately interacts with the robot.
Change in baseline parent report of child's emotion recognition | 14 weeks into treatment (at completion of intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Landa, PhD, CCC-SLP, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States